CLINICAL TRIAL: NCT03017963
Title: Safety and Tolerability of Sodium Thiosulfate in Patients Presenting With an Acute Coronary Syndrome Undergoing Coronary Angiography Via Trans-radial Approach: a Dose-escalation Study.
Brief Title: Safety and Tolerability of Sodium Thiosulfate in Patients With an ACS Undergoing CAG Via Trans-radial Approach.
Acronym: SAFE-ACS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Pim van der Harst, Prof. dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFE ACS
Record Dates: First submitted 2016-12-24; First posted 2017-01-11 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; sodium thiosulfate; maximum tolerable dose; dose-limiting toxicity
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dose-escalation cohort (Experimental): Patients are divided in 6 groups of 3 patients to receive the following intervention: 0 gram (g), 2.5 g, 5 g, 10 g, 12.5 g and 15 g of sodium thiosulfate pentahydrate (STS) intravenous. The first dose is given in 15 min immediately after inclusion at the cath-lab. In the absence of dose-limiting toxicity (DLT), a second gift of STS is given in 30 min, 6 hours later at the coronary care unit (CCU). When no DLT is observed in any of the patients after 2 gifts of the same dose an extra 3 subjects are enrolled into the next higher dose cohort. If 1 out of 3 patient develops DLT at a specific dose, an extra 3 subjects are enrolled into the same dose cohort. When more than 1 out of 6 patients develop DLT the trial will be terminated because the maximum tolerable dose (MTD) has been exceeded.
  Interventions: Drug: Sodium Thiosulfate Pentahydrate

INTERVENTIONS:
Drug: Sodium Thiosulfate Pentahydrate — Sodium Thiosulfate Pentahydrate is administered intravenously in 250 centiliters infusion fluid in two doses: first dose with an infusion rate of 16.66 milliliter (ml) per minute (min), second dose with 8.33 ml / min

SUMMARY:
The purpose of this trial is to evaluate the safety and maximum tolerable dose (MTD) of sodium thiosulfate in patients presenting with an acute coronary syndrome and treated with primary percutaneous coronary intervention (PPCI) via trans-radial approach in adjunction to standard treatment.

DETAILED DESCRIPTION:
Despite the recent advances in treatment, acute myocardial infarction (AMI) frequently results in permanent myocardial injury imposing an increased risk for adverse cardiac remodelling, diminished cardiac function and the development of heart failure. Decreased cardiac function after PPCI is associated with impaired prognosis.

Although PPCI has a tremendous benefit in AMI, not only ischemia but also reperfusion itself is considered to cause myocardial injury and cardiomyocyte death.This phenomena is referred to as "ischemia reperfusion injury" in literature and is caused by the sudden restoration of blood flow and its accompanying intracellular pH change, calcium overload, cardiomyocyte hypercontracture, myocardial inflammation, oxidative stress generation and mitochondrial permeability transition pore opening. Reducing ischemia reperfusion injury is expected to further decrease infarct size, decrease adverse cardiac remodelling and improve cardiac function as well as clinical outcome.

Hydrogen sulfide (H2S) is the third endogenous gaseous transmitter next to carbon monoxide (CO) and nitric oxide (NO) and is involved as a physiological mediator in several body organ and tissue processes. H2S is synthesized endogenously by enzymatic and non-enzymatic pathways. A non-enzymatic pathway is by the reductive reaction with thiosulfate, with pyruvate acting as a hydrogen donor. Thiosulfate itself acts as an intermediate in the sulfur metabolism of cysteine and is known as a metabolite of H2S and in that way is also able to produce H2S, especially under hypoxic conditions.

H2S has been shown to protect myocardium from ischemia reperfusion injury in various experimental animal models of ischemic heart disease; e.g. it reduces infarct size and apoptosis and attenuates cardiac function. Inhibition of leukocyte endothelial cell interactions, neutralization of reactive oxygen species (ROS) and the reduction of apoptotic signalling are the suggested as additional mechanisms underlying the cardioprotective effect of H2S in this setting.

STS, an H2S donor, is used in humans since 1933 for the treatment of cyanide intoxication and is used since the eighties for treatment of vascular calcifications in end-stage renal disease. It is also used to prevent toxicity of cisplatin treatment. More recently, studies have shown STS can delay the progression of coronary artery calcification in haemodialysis patients. The mechanism of action in these diseases is thought to be based on potential antioxidant properties of STS. In all these cases intravenous STS was used in different doses from 5 to 75 g per day. Side effects of STS include hypotension, nausea and vomiting, gastrointestinal disturbances, hypernatraemia and in 5% of hemodialysis patients metabolic acidosis occurred. Most side effects were mild and manageable.

STS administration has never been tested in the clinical setting of ACS. Cardiac catheterization via trans-radial approach has been increasingly used, instead of trans-femoral approach, resulting in fewer vascular complications, minimal risk of nerve injury and virtually no postprocedural bed rest. However, during radial approach a combination of vasodilating, blood pressure lowering and anticoagulant drugs are given to the patient (verapamil, nitroglycerin, heparin), the "radialis-cocktail". These drugs could potentially interact with STS and data regarding the safety of STS in patients with ACS treated with PCI via radial approach is lacking.

The SAFE ACS is a phase 1/2, open-label, dose-escalation study to test the hypothesis that STS, on top of standard medical treatment, can be safely administered in patients presenting with an ACS and is well-tolerated. We will use a "3+3 design" with a fixed dosing endpoint of 30 gram of STS in 2 gifts of 15 gram, based on the standard dose of 25 gram used for other indications. Additionally we will test the effect of STS treatment on oxidative stress during and after STS infusion by laboratory analysis of various oxidative stress markers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* The diagnosis ACS defined by: chest pain suggestive for myocardial ischemia for at least 30 minutes, the time from onset of the symptoms less than 24 hours before hospital admission, with (STEMI) or without (nSTEMI/uAP) an electrocardiogram (ECG) recording with ST- segment elevation of more than 0.1 millivolt (mV) in 2 or more contiguous leads;
* PCI via trans-radial approach is being considered as treatment;
* Patient is willing to cooperate with the trial during hospitalization

Exclusion Criteria:

* Known cardiomyopathy or LVEF<35%;
* History of a malignancy treated with chemo- and/or radiotherapy < 1 year;
* Systolic blood pressure under 100 mmHg or over 180 mmHg at presentation;
* Cardiogenic shock at presentation
* Sedated and/or intubated patients;
* Pregnant/breastfeeding at time of presentation
* The existence of a condition with a life expectancy of less than 1 year;
* A condition which, according to the clinical judgment of the investigator and/or treating physician, does not allow the patient to successfully participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | up to 24 hours or discharge from coronary care unit to the ward/home
  DLT defined as all-cause mortality or hemodynamic instability of significant clinical impact:
  Hemodynamic instability of significant clinical impact is defined as:
  * Systolic blood pressure <90 millimeters mercury (mmHg) for >30 min and/or
  * Catecholamines required to maintain pressure >90 mmHg during systole and
  * Signs of pulmonary congestion or elevated left-ventricular filling pressures and;
  * Signs of impaired organ perfusion with ≥1 of the following criteria:
    * Confusion;
    * Cool, clammy skin;
    * Oliguria (urine output <30 ml/h);
    * Serum-lactate >2.0 mmol/l.
  * Shock of other causes (hypovolemia, sepsis, bradycardia) are ruled out.

SECONDARY OUTCOMES:
Severe hypersensitivity/allergic reaction using a binary scale (yes/no) | up to 24 hours or discharge from coronary care unit to the ward/home
  Severe hypersensitivity/allergic reaction such as angio-edema, heavy itch/rash. Outcome measurement will assessed using a binary scale: present (yes) or absent (no)
Nausea/vomiting | up to 24 hours or discharge from coronary care unit to the ward/home
  using a 4-point Likert-scale: 0= none, 1= nauseated but able to eat and/or 1 episode of vomiting in 24 hours, 2= food intake significantly decreased and/or 2-5 episodes of vomiting in 24 hours, 3= intravenous fluids required and/or >5 episodes of vomiting in 24 hours
effect of STS on oxidative stress markers in blood | up to 12 hours
  effect of STS on oxidative stress markers in blood by laboratory analysis of free thiols in blood. Unity: µmol/l. Measurement on different timeframes, starting at T=0, to evaluate the effect of STS on free thiol levels in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Pim van der Harst, Professor, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No